CLINICAL TRIAL: NCT07200011
Title: Effect of Serum Vitamin D Levels on the Clinical and Radiographic Outcomes of Unsplinted Mandibular Implant Overdentures
Brief Title: Effect of Vitamin D on the Clinical and Radiographic of Unsplinted Mandibular Implant Overdentures
Acronym: Vit D and bone
Status: Active, not recruiting | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Rahma elhussany mohammed, Lecturer, Department of Prosthodontics, Mansoura faculty of Dentistry, Egypt, Mansoura University
Other Study IDs: R.25.07.10
Record Dates: First submitted 2025-09-03; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Vitamin D Deficiency; Implant Assesment; Radiography; Clinical and Radiographic Effect
Keywords: Vitamin D, marginal bone loss, mandibular implant overdenture, un-splinted implants, LOCATOR attachments,periapical radiographs.
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin D-deficient (<20 ng/mL): Participants with serum vitamin D <20 ng/mL
  Interventions: Other: Observational: Serum Vitamin D Levels
- Vitamin D-sufficient (≥30 ng/mL): Participants with serum vitamin D ≥30 ng/mL
  Interventions: Other: Observational: Serum Vitamin D Levels

INTERVENTIONS:
Other: Observational: Serum Vitamin D Levels — Participants' serum vitamin D levels will be measured from existing laboratory records, and radiographic images of mandibular implant overdentures will be analyzed to assess marginal bone loss. No active treatment or experimental intervention will be administered

SUMMARY:
This study investigates the effect of vitamin D on bone loss around mandibular implant overdentures. Bone levels around implants will be measured to understand how vitamin Daffect the health of implant-supported dentures. This information may help improve dental treatment outcomes

DETAILED DESCRIPTION:
Tooth loss affects patient's quality of life. The use of mandibular implant overdentures is an accepted treatment option that improves prosthesis retention, stability, and masticatory efficiency compared to conventional complete dentures.

Vitamin D plays a critical role in bone metabolism and osseointegration of dental implants. Deficiency may impair bone healing and accelerate peri-implant bone loss.

The purpose of this retrospective study is to clinically and radiographically evaluate the effect of serum vitamin D levels on peri-implant tissues in patients rehabilitated with unsplinted mandibular implant overdentures.

Patient records are screened for serum vitamin D levels, radiographs at baseline of loading and follow-up intervals ( 6 & 12 months after loading )and clinical notes.

Patients categorize into two groups based on their recorded serum vitamin D levels: group A - deficient vitamin D : < 20 ng/mL and group B - sufficient vitamin D: ≥ 30 ng/mL.

All participants rehabilitated with unsplinted, three-implant mandibular overdentures assisted by LOCATOR attachments. Minor variations in implant dimensions and positioning are accepted, provided the implants were placed in the midline and posterior regions.

All implants should be placed using a flapless surgical protocol with delayed loading protocol.

The clinical evaluation included peri-implant soft tissue parameters in patients records such as plaque index, gingival index, bleeding on probing, and probing pocket depth to monitor peri-implant health. Also, prosthesis-related factors, including stability, retention, and occlusion, were also evaluated and recorded. In addition, implant status were evaluated and recorded through mobility testing and the presence of peri-implant infection or suppuration .

Marginal bone loss (vertically and horizontally) is measured on the mesial and distal sides of each dental implant on the periapical radiographs by using the software program (Scanora light version 3.2.6; SOREDEX) calibration.

Vertical bone height (AB) is considered as the distance between the implant shoulder and the bone-to-implant contact parallel to the implant long axis. Radiographic vertical bone loss (VBL) is estimated by subtracting radiographic AB at T6 and T12 from AB at T0.

Actual VBL is calculated by multiplying the actual implant length by the radiographic VBL and dividing the result by the radiographic length of the implant to account for magnification error.

To measure the horizontal alveolar bone loss (HBL), the distance between the peri- implant bone level (C point of crest) [which is the crossing Point of the tangent to the horizontal bone crest (CD line) and the tangent to the crater-shaped defect (CB line)] and the implant at the (E Point) right angle is measured and referred to the horizontal bone level. To measure horizontal bone loss (HBL), the horizontal bone level at T6 and T12 is subtracted from T0.

Actual HBL is calculated by multiplying the actual implant diameter by the radiographic HBL and dividing the result by the radiographic diameter of the implant in order to account for magnification error.

Data are analyzed using statistical software (SPSS, version 22.0; SPSS Inc., Chicago, IL). The Shapiro-Wilk test is used to assess the normality of the bone loss data. Descriptive statistics are expressed as mean ± standard deviation. Repeated measures analysis of variance (ANOVA) is used to evaluate changes in bone loss over time, followed by the Tukey Post hoc test for pairwise comparisons between time intervals. Intergroup differences are assessed using the independent samples t test. A P value <.05 is considered statistically significant at a 95% confidence level.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 60 years.
* Patients rehabilitated with unsplinted three-implant mandibular overdentures retained by LOCATOR attachments .
* Availability of recent serum vitamin D records at determined time intervals.
* Good general health without uncontrolled systemic diseases.

Exclusion Criteria:

* Missing or incomplete patient records.
* Patients on medications known to affect bone metabolism.
* History of smoking or alcohol abuse.
* Patients with borderline serum vitamin D values (21-29 ng/mL) to avoid classification bias.
* Presence of active oral infections or untreated periodontal disease.
* Previous implant failure in the mandible.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: This retrospective study includes adult patients aged 40 to 60 years who have been rehabilitated with unsplinted three-implant mandibular overdentures retained by locator attachments. Only patients with complete clinical records, including serum vitamin D levels and adequate baseline and follow-up periapical radiographs are included. Patients with systemic diseases affecting bone metabolism, history of smoking or alcohol abuse, or medications known to influence bone healing are excluded. The study population are stratified based on serum vitamin D levels into two groups: deficient (<20 ng/mL) and sufficient (≥30 ng/mL)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum vitamin D levels and radiographic marginal bone loss around unsplinted mandibular implant overdentures | Baseline (prosthetic loading), 6 months, 12 months after loading (T0,T6,T12)
  Marginal bone loss vertically (VBL) and horizontally (HBL) around each unsplinted mandibular dental implant are measured on standardized digital periapical radiographs using Scanora Light software (mm).
  Serum vitamin D levels (ng/mL) are obtained from patient records. The correlation between serum vitamin D concentration and marginal bone loss will be analyzed.

SECONDARY OUTCOMES:
Clinical & peri-implant outcomes of unsplinted mandibular implant overdentures Peri-implant soft tissue health: plaque index , gingival index, bleeding on probing | Baseline (prosthetic loading), 6 months, 12 months after loading T0, T6,T12
  Clinical and peri-implant parameters are assessed from patient avilable records and clinical examinations. Peri-implant soft tissue health were evaluated in patients records by using plaque index , gingival index , bleeding on probing.
  Unit of Measure / Measurement Tool:
  Plaque Index % (PI%) (Patient chart records) Gingival Index % (GI %) (Patient chart records) Bleeding on Probing % (BOP% ) (Patient chart records)
Clinical and peri-implant parameters are assessed from patient avilable records and clinical examinations: probing pocket depth | Baseline (prosthetic loading), 6 months, 12 months after loading T0, T6,T12
  Clinical and peri-implant parameters are assessed from patient avilable records and clinical examinations. Peri-implant probing pocket depth was evaluated in patients records peridontal probe.
  Unit of Measure / Measurement Tool:
  Probing Pocket Depth (mm) (Patient chart records)
Implant status including mobility and presence of peri-implant infection or suppuration were also evaluated and recorded in all patients data. | Baseline (prosthetic loading), 6 months, 12 months after loading T0, T6,T12
  Mobility Unit: Qualitative (Present / Absent) Clinical significance: presence of mobility indicates loss of osseointegration and implant failure.
  Peri-implant infection / suppuration Unit: Qualitative (Present / Absent) Recorded when signs of infection (e.g., purulent exudate, swelling, erythema) were detected upon probing or palpation.
Prosthesis-related factors, including stability, retention, and occlusion, were assessed clinically. | Baseline (prosthetic loading), 6 months, 12 months after loading T0, T6,T12
  Stability Unit: Qualitative (Good / Poor) Refers to absence of rocking or movement of the overdenture under functional load.
  Retention Unit: Qualitative (Adequate / Inadequate) Determined by resistance of the overdenture to vertical dislodgement when gentle pulling is applied.
  Occlusion Unit: Qualitative (Acceptable / Unacceptable) Evaluated based on even bilateral contacts, absence of premature contacts, and proper centric occlusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
This study is a retrospective observational study using existing patient records. Individual participant data will not be shared to protect patient confidentiality and privacy, and due to restrictions in accessing historical medical records

REFERENCES:
- See also: Direct procedure for connecting a mandibular implant-retained overdenture with ball attachments — https://pubmed.ncbi.nlm.nih.gov/15507918/
- See also: A within-subject clinical trial on the conversion of mandibular two-implant to three-implant overdenture: Patient-centered outcomes and willingness to pay — https://pubmed.ncbi.nlm.nih.gov/30681193/
- See also: Comparison of masticatory efficiency, patient satisfaction for single, two, and three implants supported overdenture in the same patient: A pilot study — https://pubmed.ncbi.nlm.nih.gov/27141169/
- See also: Clinical and radiographic evaluation of three-implant-retained mandibular overdentures: a 3-year retrospective study — https://pubmed.ncbi.nlm.nih.gov/21909496/
- See also: Vitamin D and intestinal calcium absorption — https://pubmed.ncbi.nlm.nih.gov/21664413/
- See also: Is Low Serum Vitamin D Associated with Early Dental Implant Failure? A Retrospective Evaluation on 1625 Implants Placed in 822 Patients — https://pubmed.ncbi.nlm.nih.gov/27738389/
- See also: Correlation of Serum Vitamin D with Crestal Bone Level in Dental Implant Patients Using CBCT: A Clinical Retrospective Study — https://pubmed.ncbi.nlm.nih.gov/37622616/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT07200011/Prot_SAP_ICF_000.pdf